CLINICAL TRIAL: NCT02010203
Title: Phase 1/2, Placebo-Controlled, Randomized Study to Evaluate the Safety, Immune Response & Clinical Activity of HS-410 in Patients With Non-Muscle Invasive Bladder Cancer Who Have Undergone Transurethral Resection of Bladder Tumor (TURBT)
Brief Title: A Phase 1/2 Study of HS-410 in Patients With Non-Muscle Invasive Bladder Cancer After TURBT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inability to accrue due to changing treatment landscape (PD-1 approvals)
Sponsor: Heat Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS410-101
Record Dates: First submitted 2013-12-05; First posted 2013-12-12 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Bladder Cancer
Keywords: TURBT; Bladder; Cancer; GP96; Vaccine; Immunotherapy; Heat Biologics; BCG; Bacillus Calmette-Guerin; Bacillus Calmette-Guérin
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms | interventions — BCG Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Phase I: HS-410 Low Dose (Experimental): In the open label Phase 1 portion, HS-410 is given as 1*10^6 cells per dose for 12 weekly injections followed by 3 monthly injections.
  Interventions: Biological: HS-410
- Phase II: HS-410 Low-Dose Plus BCG (Experimental): In the Phase 2 portion, HS-410 is given as 1*10^6 cells per dose weekly for 6 weeks in combination with BCG, followed by 6 weeks of HS-410 alone, and then 3 courses of three once-weekly doses of HS-410 in combination with BCG.
  Interventions: Biological: HS-410; Biological: BCG
- Phase II: High-Dose HS-410 Plus BCG (Experimental): In the Phase 2 portion, HS-410 is given as 1*10^7 cells per dose weekly for 6 weeks in combination with BCG, followed by 6 weeks of HS-410 alone, and then 3 courses of three once-weekly doses of HS-410 in combination with BCG.
  Interventions: Biological: HS-410; Biological: BCG
- Phase II: Placebo Plus BCG (Placebo Comparator): In the Phase 2 portion, a placebo is given weekly for 6 weeks in combination with BCG, followed by 6 weeks of placebo alone, and then 3 courses of three once-weekly doses of placebo in combination with BCG.
  Interventions: Biological: Placebo; Biological: BCG
- Phase II: High-Dose HS-410 (Experimental): In the Phase II portion, if patients will not receive BCG, HS-410 is given as 1*10^7 cells per dose weekly for 12 weeks, and then 3 courses of three once-weekly doses of HS-410.
  Interventions: Biological: HS-410

INTERVENTIONS:
Biological: HS-410 — Vaccine derived from irradiated cancer cells genetically engineered to continually secrete gp96
  Arms: Phase I: HS-410 Low Dose; Phase II: HS-410 Low-Dose Plus BCG; Phase II: High-Dose HS-410; Phase II: High-Dose HS-410 Plus BCG
Biological: Placebo — Injection containing sterile solution but no cells
  Arms: Phase II: Placebo Plus BCG
Biological: BCG — Vaccine derived from a live bacterium
  Other Names: Bacillus Calmette-Guerin
  Arms: Phase II: HS-410 Low-Dose Plus BCG; Phase II: High-Dose HS-410 Plus BCG; Phase II: Placebo Plus BCG

SUMMARY:
Phase I/II study: Phase 1 is an open-label, safety study, patients who previously received 3-6 instillations of weekly intravesical Bacillus Calmette-Guerin (BCG) induction therapy (as standard of care) followed by low dose intradermal (1*10^6 cells) HS-410 monotherapy. Phase 2, patients will be randomized to one of three blinded (physician-patient), placebo-controlled groups and receive either intradermal placebo or low dose (1*10^6 cells) or high dose (1*10^7 cells) vesigenurtacel-L in combination with induction and maintenance intravesical BCG. Patients who do not receive BCG will be enrolled into an open-label, non-randomized group receiving high dose (1*10^7 cells) intradermal HS-410 monotherapy.

DETAILED DESCRIPTION:
This study is a two part study: Phase I and Phase II. The Phase 1 portion is an open-label, safety study. Patients will have previously received 3-6 instillations of weekly intravesical Bacillus Calmette-Guerin (BCG) induction therapy (as standard of care) followed by low dose intradermal (1*10^6 cells) HS-410 monotherapy. In Phase 2, patients will be assigned to treatment groups based on whether they will receive induction BCG in the typical post-TURBT window. If the investigator plans to administer BCG, patients will be randomized to one of three blinded (physician-patient), placebo-controlled groups and receive either intradermal placebo or low dose (1*10^6 cells) or high dose (1*10^7 cells) vesigenurtacel-L in combination with induction and maintenance intravesical BCG. If patients will not receive BCG, they will be enrolled into an open-label, non-randomized group and receive high dose (1*10^7 cells) intradermal HS-410 monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-muscle invasive bladder cancer [Ta, T1 or Tis (CIS)] that has been removed by transurethral resection
* Either: (i) high-risk disease, defined as T1 and/or high-grade and/or CIS or (ii) intermediate-risk disease, defined as Ta low-grade with at least 3 of the following 4 risk factors: multiple tumors, tumor size > 3cm, early recurrence (<1 year from previous staging procedure), or recurrence with a frequency of more than once in any 12 month period
* Not have received bacillus Calmette-Guérin (BCG) or have completed previous BCG treatment > 12 months prior to the baseline staging procedure.
* Phase 2 Arms 1-3: Suitable to receive a 6-week course of BCG in the adjuvant setting within 6 weeks following TURBT. Phase 2 Arm 4: Suitable for monotherapy vaccine administration post-TURBT. For Phase 1 only: Has previously received 3-6 weekly doses of BCG.
* Adequate laboratory parameters

Exclusion Criteria:

* Human immunodeficiency virus (HIV) infection or immunodeficiency disorders, either primary or acquired
* Infections or intercurrent illness requiring active therapy
* Any condition requiring active steroid or other immunosuppressive therapy
* Active malignancies within the past 12 months except negligible risk of metastasis or death treated with expected curative outcome.
* Prostate pelvic radiation within the past 12 months
* Significant cardiac impairment
* Current alcohol or chemical abuse, or mental or psychiatric condition precluding protocol compliance
* Pregnant or nursing
* Allergy to soy, egg, or peanut products
* Receiving another investigational agent (30 day wash-out required prior to first dose)
* Neo-adjuvant therapy prior to baseline staging procedures for the current occurrence of non-muscle invasive bladder cancer
* Prior treatment with a cancer vaccine for this indication
* Prior vaccination with BCG for tuberculosis disease
* Prior splenectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-12; Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Steinberg, MD, Principal Investigator — University of Chicago
Locations (19):
- United States (19):
  - University of California at Los Angeles, Los Angeles, California
  - Skyline Urology, Sherman Oaks, California
  - Skyline Urology, Torrance, California
  - Urology Center of Colorado, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - First Urology, Jeffersonville, Indiana
  - Horizon Oncology Research, Lafayette, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - University of Massachusetts, Worcester, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology of North Texas, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Urology of Virginia, Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase I: HS-410 Low Dose | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Started | 10 | 26 | 26 | 26 | 16
Completed | 10 | 17 | 16 | 23 | 3
Not Completed | 0 | 9 | 10 | 3 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: HS-410 Low Dose | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410 | Total
Number analyzed (Participants) | 10 | 26 | 26 | 26 | 16 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 7 | 12 | 6 | 1 | 27
  >=65 years | 9 | 19 | 14 | 20 | 15 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (7.495) | 70.5 (11.176) | 68.58 (11.518) | 70.58 (9.047) | 72.50 (9.784) | 70.60 (10.172)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 5 | 6 | 3 | 18
  Male | 9 | 23 | 21 | 20 | 13 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 2 | 0 | 5
  Not Hispanic or Latino | 10 | 25 | 24 | 24 | 16 | 99
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 0 | 2
  White | 10 | 26 | 25 | 23 | 16 | 100
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 26 | 26 | 26 | 16 | 104

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Safety and Tolerability
Description: To evaluate the safety and tolerability of vesigenurtacel-L
Time Frame: Up to 3 years.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I: HS-410 Low Dose: HS-410 is given as 1*10^6 cells per dose for 12 weekly injections followed by 3 monthly injections.
Arm/Group | Phase I: HS-410 Low Dose
Number analyzed (Participants) | 10
Participants
  Gastrointestinal Disorders | 3
  General Disorders & Administration Site Conditions | 5
  Musculoskeletal & Connective Tissue Disorders | 1

2. Primary Outcome: Phase 2: 1-year Disease-Free Survival
Description: Arm 1, 2, 3: 1-year DFS in patients with NMIBC treated with BCG in combination with blinded study product (one of two doses of vesigenurtacel-L or placebo) Arm 4: 1-year DFS in patients with NMIBC treat1fv 9 with high dose vesigenurtacel-L monotherapy
  One-year disease-free survival will be defined as the proportion of patients who are free from recurrent disease, progressive disease, and alive one year after the date of randomization/treatment assignment
Time Frame: One year
Population: Phase I is not applicable since the Outcome Measure is solely for Phase II; as pre-specified, only Phase II data would be collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Number analyzed (Participants) | 26 | 26 | 26 | 16
Participants | 7 | 9 | 6 | 12

3. Secondary Outcome: Proportion of Patients With Recurrence at 3, 6, 12, 18, and 24 Months
Description: Evaluate the proportion of patients with recurrence at 3, 6, 12, 18, and 24 months
Time Frame: Up to 2 years
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Number analyzed (Participants) | 26 | 26 | 26 | 16
participants
  3 months | 22 | 19 | 23 | 14
  6 months | 19 | 19 | 22 | 9
  12 months | 18 | 17 | 21 | 4
  18 months | 18 | 16 | 15 | 2
  24 months | 14 | 14 | 12 | 1

4. Secondary Outcome: Proportion of Patients With Progressive Disease at 3, 6, 12, 18, and 24 Months
Description: Evaluate the proportion of patients with progressive disease at 3, 6, 12, 18, and 24
Time Frame: Up to 2 years
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Number analyzed (Participants) | 26 | 26 | 26 | 16
participants
  3 Months | 1 | 1 | 0 | 0
  6 Months | 2 | 3 | 0 | 3
  12 Months | 2 | 3 | 1 | 3
  18 Months | 2 | 3 | 2 | 4
  24 Months | 2 | 3 | 2 | 4

5. Secondary Outcome: Disease-free Survival at 3, 6, 18, and 24 Months
Description: Evaluate Disease Free Survival at 3, 6, 18 and 24 months
Time Frame: Up to 2 years
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Number analyzed (Participants) | 26 | 26 | 26 | 16
participants
  3 months | 22 | 19 | 23 | 14
  6 months | 19 | 19 | 22 | 9
  12 months | 18 | 17 | 21 | 4
  18 months | 17 | 16 | 15 | 2
  24 months | 13 | 14 | 12 | 1

6. Secondary Outcome: Overall Disease-free Survival
Description: Evaluate overall Disease Free Survival
Time Frame: Up to 3 years
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Number analyzed (Participants) | 26 | 26 | 26 | 16
participants | 18 | 17 | 18 | 3

7. Secondary Outcome: Overall Survival, Expressed as the Number of Participants Alive
Description: Evaluate overall survival (OS)
Time Frame: Up to 3 years
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Number analyzed (Participants) | 26 | 26 | 26 | 16
participants | 26 | 26 | 26 | 16

8. Secondary Outcome: Proportion of Patients Undergoing Repeat Transurethral Resection of Bladder Tumor (TURBT) by 12 and 24 Months
Time Frame: Up to 2 years
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG
Number analyzed (Participants) | 26 | 26 | 26
participants
  12 Month | 8 | 6 | 10
  24 Months | 8 | 7 | 11

9. Secondary Outcome: Proportion of Patients Undergoing Cystectomy by 12 and 24 Months
Description: Evaluate the proportion of patients undergoing cystectomy by 12 and 24 months from randomization
Time Frame: Up to 2 years
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Number analyzed (Participants) | 26 | 26 | 26 | 16
participants
  12 Months | 0 | 0 | 0 | 1
  24 Months | 1 | 0 | 0 | 1

10. Secondary Outcome: Immunologic Response of PBMCs Via Intracellular Cytokine Staining (ICS) by Flow Cytometry and/or Enzyme-linked Immunosorbent Spot (ELISPOT) on CD8+ Cells After HS-410 Vaccination as Compared to Baseline.
Description: Evaluate the proportion of patients with immunologic response of peripheral blood mononuclear cells (PBMCs) via intracellular cytokine staining (ICS) by flow cytometry and/or ELISPOT on CD8+ cells following vesigenurtacel-L vaccination
Time Frame: Up to 2 years
Population: Data were not collected as pre-specified in Outcome Measure 10 due to study termination by the Sponsor.
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Immunologic Response of Peripheral Blood Mononuclear Cells (PBMCs) and Stimulation Analysis Via ICS in Baseline and Post-treatment Biopsies, if Clinically Indicated
Description: Evaluate immunologic response of PBMCs (analysis of surface markers, CD3, CD4, CD8, CD19, CD25, CD45, CD56, FoxP3, and degranulation) and stimulation analysis via ICS of interferon gamma (IFNγ) and granzyme B (gzB)
Time Frame: Up to 3 years
Population: Data were not collected as pre-specified in Outcome Measure 11 due to study termination by the Sponsor.
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Total PBMC Counts by Flow Cytometry
Description: Evaluate total PBMC counts by flow cytometry, including lymphocyte subsets (B cells, helper T-cells, cytotoxic T-cells, natural killer (NK) cells and T-reg)
Time Frame: Up to 3 years
Population: Data were not collected as pre-specified in Outcome Measure 12 due to study termination by the Sponsor.
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Tumor Antigen Expression
Description: Evaluation of pre-treatment tumor tissue for antigen expression
Time Frame: At screening
Population: Data were not collected as pre-specified in Outcome Measure 13 due to study termination by the Sponsor.
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Tumor Infiltrating Lymphocytes (TILs)
Description: Evaluation of tumor tissue obtained from repeat biopsy, if clinically indicated, for presence of TILs
Time Frame: Up to 3 years
Population: Data were not collected as pre-specified in Outcome Measure 14 due to study termination by the Sponsor.
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: T Cell Receptor Sequencing of Peripheral Blood T Cells Before and During Treatment
Description: Evaluation of tumor tissue obtained from repeat biopsy, if clinically indicated, for presence of TILs, T cell receptor sequencing of peripheral blood T cells before and during the course of treatment.
Time Frame: Up to 2 years
Population: Data were not collected as pre-specified in Outcome Measure 15 due to study termination by the Sponsor.
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Safety of the Combination of the HS-410 and BCG
Description: Phase 2 only Evaluate the safety of the combination of vesigenurtacel-L and BCG
Time Frame: Up to 1 year
Population: Data were not collected as pre-specified in Outcome Measure 16 due to study termination by the Sponsor.
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Safety of the High Dose HS-410 Monotherapy
Description: Phase 2 only Evaluate the safety of high dose vesigenurtacel-L monotherapy
Time Frame: Up to 3 years.
Population: Data were not collected as pre-specified in Outcome Measure 17 due to study termination by the Sponsor.
Arm/Group | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were defined as all reported events with a start date on or after Study Day 1. All AEs were collected through 30 days post last dose, up to 3 years.
Arm/Group | Phase I: HS-410 Low Dose | Phase II: HS-410 Low-Dose Plus BCG | Phase II: High-Dose HS-410 Plus BCG | Phase II: Placebo Plus BCG | Phase II: High-Dose HS-410
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/26 | 0/26 | 0/26 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/10 | 8/26 | 4/26 | 1/26 | 2/16
Other Adverse Events (participants affected / at risk) | 7/10 | 24/26 | 19/26 | 20/26 | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: HS-410 Low Dose (N=10) | Phase II: HS-410 Low-Dose Plus BCG (N=26) | Phase II: High-Dose HS-410 Plus BCG (N=26) | Phase II: Placebo Plus BCG (N=26) | Phase II: High-Dose HS-410 (N=16)
Cystoprostatectomy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate Cancer (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — Mycotic Aneurysm; Disseminated BCG Mycotic Aneurysm
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — of Larynx
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Priapism (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder Perforation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: HS-410 Low Dose (N=10) | Phase II: HS-410 Low-Dose Plus BCG (N=26) | Phase II: High-Dose HS-410 Plus BCG (N=26) | Phase II: Placebo Plus BCG (N=26) | Phase II: High-Dose HS-410 (N=16)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (7) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 5 (8) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 5 (10) | 4 (5) | 3 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 10 (14) | 6 (11) | 4 (4) | 3 (3)
Influenza Like Illness (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 5 (7) | 3 (3) | 3 (4) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 8 (8) | 3 (4) | 6 (7) | 0 (0)
Blood Urine Present (Investigations) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Hematocrit Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White Blood Cell Count Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 3 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (4) | 0 (0)
Cerebrovascular Disorder (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (4) | 2 (2) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Bladder Perforation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder Spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (10) | 6 (18) | 9 (11) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 6 (9) | 5 (13) | 3 (4) | 0 (0)
Lower Urinary Tract Symptoms (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Micturition Urgency (Renal and urinary disorders) | 0 (0) | 5 (5) | 4 (19) | 3 (6) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 5 (6) | 4 (18) | 3 (5) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breast Tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (4) | 2 (2) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (5) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Injection Site Pain (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperadrenalism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder Spasm (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-02-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT02010203/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/03/NCT02010203/SAP_001.pdf